CLINICAL TRIAL: NCT00175305
Title: Effect of Somatostatin on Ghrelin Concentrations, Food Seeking Behaviour and Weight in Patients With Prader-Willi Syndrome
Brief Title: Prader-Willi Syndrome and Appetite
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C04-0007; W04-0007
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Hyperphagia; Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; Somatostatin; Ghrelin; Obesity; Hyperphagia; Hyperphagia in Prader-Willi syndrome
MeSH Terms: conditions — Hyperphagia; Prader-Willi Syndrome; Obesity

INTERVENTIONS:
Drug: Sandostatin LAR

SUMMARY:
Excessive weight gain is a cardinal feature of Prader-Willi syndrome (PWS) for which there is presently no effective treatment. It is caused by increased appetite, decreased perception of satiety and obsessive and compulsive behaviour towards food. Ghrelin is a powerful appetite-stimulating hormone. Patients with PWS have markedly elevated ghrelin levels, suggesting that it may be responsible for the increased food intake. The goal of the study is to determine whether treatment with somatostatin (Sandostatin), a hormone that inhibits ghrelin, is an effective treatment for the prevention and treatment of weight excess in patients with PWS.

DETAILED DESCRIPTION:
Prader-Willi Syndrome and Obesity:

Prader-Willi syndrome (PWS) is a genetic disorder occurring in 1/10,000 to 1/15,000 live births. Clinical characteristics include neonatal and infantile central hypotonia with feeding problems and poor weight gain followed after 1-3 years by hyperphagia and excessive weight gain. Patients also have characteristic facial features, short stature (possibly due to growth hormone [GH] deficiency of hypothalamic origin), hypogonadism, increased pain threshold, global developmental delay and variable mental retardation.

Obesity is clearly one of the cardinal features of PWS. It can result in tremendous distress for both the parents and the affected child and is a significant health problem with complications that include hypertension, sleep apneas and diabetes. More than 1/3 of patients with PWS weigh more than 200% of their ideal body weight. Obesity is thought to result mainly from hyperphagia, persistent hunger with increased caloric intake, decreased perception of satiety and obsessive and compulsive behaviours that are primarily food related. Decreased physical activity associated with hypotonia and/or decreased energy expenditure is also thought to play a role in the pathophysiology of obesity.

The treatment of obesity in PWS is very difficult and requires constant involvement of the parents or caregivers with establishment of rigid structures around the young patient: increased physical activity, hiding food, locking fridges etc. Recently, studies on the effects of growth hormone (GH) treatment (now an approved indication in most patients with PWS in the US irrespective of their GH status) on body composition in PWS have been performed. While GH, among other favourable effects, significantly improves body composition (increased lean mass and decreased fat mass), the long-term effects on body mass index are modest and variable.

Thus, obesity is clearly one of the greatest challenges faced by parents of patients with PWS and treatment modalities are presently not successful.

Ghrelin:

Ghrelin is a recently discovered peptide that stimulates appetite and GH secretion. Ghrelin increases with fasting and decreases following a meal, and is thought to play a role in meal initiation in humans. In obese adult and young patients (without PWS), ghrelin is decreased compared to control, lean subjects suggesting that it does not play a causal role in the development of obesity. In contrast, PWS patients are characterized by extremely high circulating ghrelin levels (3 to 10 times higher compared to controls). The mechanisms underlying ghrelin increase in PWS are unclear. The gene encoding ghrelin is located on chromosome 3 in humans while PWS is associated with the functional loss of paternally expressed genes located on chromosome 15 (most patients affected with PWS present with a deletion in the area of 15q11-13 [70%] or a uniparental disomy for maternal chromosome 15 [30%]). A logical hypothesis is that these missing genes may be part of a pathway regulating ghrelin expression.

Thus, the elevated ghrelin concentrations observed in PWS at the very least raise the possibility that ghrelin may play an etiological role in the food-seeking behaviour reported in these patients. In support of this hypothesis, a significant correlation between hunger sensation and ghrelin concentrations has recently been reported in a combined group of 6 lean controls and 7 patients with PWS.

Somatostatin and Somatostatin Analogues:

Somatostatin is a hormone that circulates under 2 main forms: a 14 amino acid peptide (SST-14, mainly in the brain, including the hypothalamus) and a 28 amino acid peptide (SST-28, mainly in the gastrointestinal tract). Somatostatin inhibits GH and insulin secretion. Somatostatin is also a powerful regulator of gastric activity that decreases gastrin release, acid output and gastric motility.

The somatostatin analogue octreotide (Sandostatin®, Novartis) contains 8 amino acids and is very similar to SST-14. It is an effective treatment of neonatal hyperinsulinism (a condition characterized by excessive and inappropriate secretion of insulin that causes severe hypoglycemia in infants) and acromegaly (a condition characterized by excessive GH production by the pituitary). Sandostatin LAR® is a recent long-acting analogue of somatostatin that is used for the treatment of acromegaly and less often in children's hyperinsulinism.

Sandostatin LAR® therapy may be associated with significant side-effects):

* Reduction of bile production and gallbladder contractility and increased risk of cholesterol gallstones. However, these tend to resolve either spontaneously when therapy is discontinued or with ursodiol despite remaining on therapy. Therefore, gallbladder ultrasound is part of the routine follow-up of all patients receiving octreotide for prolonged periods.
* Decreased height velocity secondary to inhibition of GH secretion. This effect is variable in intensity but present and will need to be taken into account in case of prolonged octreotide treatment. In the proposed study, 12 weeks of octreotide treatment are not expected to have a significant long-term effect on longitudinal growth. Octreotide should not interfere with GH action in PWS subjects receiving concomitant exogenous human GH.
* Glucose intolerance. Prolonged octreotide treatment has been associated with impaired glucose tolerance secondary to a decrease in insulin secretion. However, when octreotide treatment results in weight loss, an improvement in glucose tolerance is observed. Therefore, parameters reflecting glucose tolerance must be followed as part of Sandostatin LAR® therapy.

Other side effects include nausea, abdominal cramps, diarrhea and flatulence that usually subside after 2 weeks of treatment.

Effect of Somatostatin Analogues on Ghrelin and Weight Gain:

Somatostatin has been shown to decrease ghrelin concentrations in normal subjects as well as in patients with PWS and with acromegaly. In nine lean young men, continuous SC infusion of octreotide (600 microg/24 hours) caused a 50% decrease in ghrelin concentrations. In patients with PWS, using the dose of 5 microg Sandostatin/kg body weight, SC, three times a day, Hacqq et al observed a 67% drop in ghrelin concentrations. The study was of short duration (1 week) but the results suggest that somatostatin may indeed be helpful in decreasing ghrelin concentrations in patients with PWS. There were no complications. In adults with acromegaly (aged 25-59 years, mean BMI 28.9 kg/m2), fasting ghrelin concentrations decreased in all patients (mean 54%, range 30-74) following treatment with Sandostatin LAR® (10 to 30 mg/4-6 weeks) for 3-29 months. Finally, Lustig et al reported the effects of daily injections of octreotide for 6 months in a group of children with severe hypothalamic obesity due to brain tumor treatment and/or cranial irradiation. They observed that the weight gain in octreotide-treated patients was minimal (+ 1.2 kg/6 mo) compared to the placebo group (+ 9.2 kg/6 mo). Bile sludging and/or gallstones were observed in 44% of the patients but resolved with ursodiol therapy. Ghrelin concentrations were not measured in that study.

Thus, somatostatin analogues cause a marked decrease in ghrelin concentrations in control subjects as well as in patients with PWS. Whether they are associated with a sustained decrease in ghrelin concentrations and whether the decrease in ghrelin is associated with a decrease in appetite is unknown and will be studied in the present project.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Prader-Willi syndrome, confirmed by genetic testing

Ages: 10 Years to 17 Years | Sex: All
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2004-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Changes in ghrelin concentrations during a test meal | 8 to 10 AM

SECONDARY OUTCOMES:
Change in weight, behaviour and food intake

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Chanoine, MD, Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada